CLINICAL TRIAL: NCT06361771
Title: Evaluation of Invisible Preparation Behaviors of Middle and High School Students in Sports Facilities
Brief Title: Evaluation of Invisible Preparation Behaviors of Middle and High School Students in Sports Facilities (PRICELESS)
Acronym: PRICELESS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0079 - PRICELESS
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Sports Injury; Prevention; Training; Hydration; Nutrition; Sleep; Mental Health; Physical Well-Being
MeSH Terms: conditions — Athletic Injuries; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators define the Invisible Preparation (IP) as the set of health behaviors that young athletes implement, on their own, to optimize their health and performances. This includes sleep, nutrition and hydration, physical well-being (injuries prevention) and mental well-being. If some studies have reported a lack of compliance in young athletes regarding sleep and hydration recommendations, the literature is poor in this field.

The CMS (Brest Metropolitan Area Sports Medicine Centre, France) aims at preserving the health of young athletes. Prior to their medical examination, the patients will be asked, all along the year 2024, to fill out a form that question them about their health behaviors in the four areas of the IP.

Under the direction of the Brest University Hospital, PRICELESS (Invisible Preparation of Middle and High School Students in Sports Institutions) study will try, based on their answers, to estimate the proportion of young athletes who declare adopting the health behaviors recommended in the IP.

ELIGIBILITY:
Inclusion Criteria:

* Middle and High School students
* Being part of a Sports Institution (Club, Sport Section at School, Local Training Institution, or Elite Training Institution)
* Absence of opposition from the patients or their legal representatives

Exclusion Criteria:

* Primary School and College students
* Refusal to participate
* Significant mental or psychological disability, making it impossible to obtain reliable answers

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Middle and High School students who are part of a Sports Institution (Club, Sport Section at School, Local Training Institution, or Elite Training Institution), in Brest, Brittany, France, and its surroundings
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
The proportion of teenagers who declare adopting the health behaviors recommended in the four areas of the Invisible Preparation. | january - december 2024

SECONDARY OUTCOMES:
The proportion of girls who declare adopting these behaviors, compared to the proportion in boys. | january - december 2024
The proportion of Middle School students who declare adopting these behaviors, compared to the proportion in High School students. | january - december 2024
The proportion of young athletes practicing an intensive sporting activity (10 hours or more per week), compared to the proportion in young athletes practicing a non-intensive sporting activity (less than 10 hours per week). | january - december 2024
The proportion of young athletes with disabilities who declare adopting these behaviors, compared to the proportion in young athletes without disabilities. | january - december 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement